CLINICAL TRIAL: NCT03082287
Title: ALPCO Calprotectin ELISA - Measurement of Calprotectin Levels in Human Stool
Status: Completed | Type: Observational
Sponsor: American Laboratory Products Company (Industry)
Collaborators: MDC Associates, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALPCOCAL
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- IBD: Adult subjects diagnosed with IBD via endoscopy and histological findings.
  Interventions: Device: Fecal Calprotectin Level
- IBS: Adult subjects with IBS as per the Rome IV criteria.
  Interventions: Device: Fecal Calprotectin Level
- Other GI Disorders: Adult subjects with gastrointestinal disorders not meeting the Rome IV criteria or IBD diagnosis.
  Interventions: Device: Fecal Calprotectin Level
- Healthy Subjects: Adult subjects without any gastrointestinal complaints.
  Interventions: Device: Fecal Calprotectin Level

INTERVENTIONS:
Device: Fecal Calprotectin Level — Measurement of calprotectin in feces

SUMMARY:
The ALPCO Calprotectin ELISA is an in vitro diagnostic test intended to quantitatively measure concentrations of fecal calprotectin in human stool samples. Calprotectin is a protein biomarker of mucosal inflammation. Measurement of calprotectin can aid in the diagnosis of Inflammatory Bowel Diseases (IBD), specifically Crohn's Disease (CD) and Ulcerative Colitis (UC), as well as aid in the differentiation of IBD from Irritable Bowel Syndrome (IBS) when used in conjunction with other diagnostic testing and the total clinical picture. This study will estimate the predictive values of a negative (NPV) and positive (PPV) test by utilizing the assay outcomes of the ALPCO Calprotectin ELISA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (IBD or IBS subjects):

* >18 years of age
* Patient must present with signs and symptoms of IBS or IBD
* Patient must be scheduled for a colonoscopy
* All results of the colonoscopy including histology must be provided to study site and sponsor.
* Medical Chart review may be required to confirm diagnosis of IBS or IBD
* Patient must not have taken NSAIDs for at least 2 weeks prior to participating in the study. Patients may be advised of the study and if report taking NSAIDS may be enrolled in the study after the patient has stopped use of NSAIDS for a minimum of 2 weeks.
* For normal patient population - study participants must present with no signs or symptoms of IBS or IBD, must not have taken NSAIDs for at least a period of 2 weeks and must be willing to provide a stool sample.
* Sample must be collected at least 2-3 days prior to colonoscopy

Inclusion Criteria (normal subjects):

* Male or female, ≥18 years of age.
* No abdominal complaints and no history of IBS, IBD, or other chronic intestinal disorder, confirmed by medical history and physical examination at enrollment.
* May have undergone colonoscopy with negative findings within the past 1 month or may have no recent colonoscopy, but scheduled for routine screening colonoscopy.
* Able to understand the study and the task required, and sign the ICF.

Exclusion Criteria:

Exclusion Criteria (IBD or IBS Subjects):

* patient under the age of 18
* Patient taking NSAIDs
* Patients not presenting with signs or symptoms of IBS or IBD with the exception of 100 normal patients to be included in the study. Fifty (50) presenting for routine colonoscopy and 50 patients presenting with no disease symptoms and not scheduled for a colonoscopy.
* Patients not scheduled to have an colonoscopy unless enrolled in the study as normal population

Exclusion Criteria (normal subjects):

* Unable or unwilling to provide a stool specimen.
* Have taken protein pump inhibitors (PPIs) or H2-receptor antagonists for control of upper GI disease within the previous 2 weeks.
* Have taken NSAIDs (including aspirin) on within 2 weeks of study enrollment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals that presents with symptoms of IBS/IBD and otherwise healthy subjects
Sampling Method: Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
In vitro diagnostic value of Calprotectin | Through study completion, up to 52 weeks.
  Value of calprotectin measurement in the ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Fran White, Study Director — MDC Associates
Locations (1):
- ALPCO, Salem, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No